CLINICAL TRIAL: NCT00958451
Title: Response of Secondary Hyperparathyroidism to Paricalcitol Versus Ergocalciferol in Patients With Stage 3 and 4 Chronic Kidney Disease With Vitamin D Deficiency: a Randomized Controlled Trial
Brief Title: Vitamin D Deficiency in Chronic Kidney Disease (CKD) Patients
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Salem Veterans Affairs Medical Center (U.S. Federal Agency)
Collaborators: Abbott (Industry)
Responsible Party: Csaba P. Kovesdy, M.D., Salem VAMC
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CK0023
Record Dates: First submitted 2009-08-11; First posted 2009-08-13 (Estimated); Last update posted 2011-03-24 (Estimated); Status verified 2009-08

CONDITIONS: Secondary Hyperparathyroidism; Chronic Kidney Disease
Keywords: Calcium; Vitamin D deficiency; Chronic Kidney disease
MeSH Terms: conditions — Hyperparathyroidism, Secondary; Renal Insufficiency, Chronic; Vitamin D Deficiency | interventions — paricalcitol; Ergocalciferols

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Paricalcitol (Active Comparator): Arm 1: 40 patients will be assigned to paricalcitol treatment group. Patients will be randomized once they meet inclusion and exclusion criteria. If patients are not on any vitamin D treatment when enrolled, they will have 2 screening visits before randomization. Screening visits will consist of a physical exam and lab tests to measure Vitamin D, calcium, iPTH, and safety profile. Patients on vitamin D treatment prior to study will have a minimum 4 week washout period before screening tests. Patients' Lean Body Mass and Aortic Blood Pressure and pulse wave velocity will be measured before dosing. Cardiovascular markers will be checked throughout the study. Patients will be monitored monthly after starting study treatment. Total treatment period: 4 months.
  Interventions: Drug: Paricalcitol; Drug: Ergocalciferol
- Ergocalciferol (Active Comparator): Arm 2: 40 patients will be assigned to the Ergocalciferol treatment group. Patients will be randomized once they meet inclusion and exclusion criteria. If patients are not on any vitamin D treatment when enrolled, they will have 2 screening visits before randomization. Screening visits will consist of a physical exam and lab tests to measure Vitamin D, calcium, iPTH, and safety profile. Patients on vitamin D treatment prior to study will have a minimum 4 week washout period before screening tests. Patients' Lean Body Mass and Aortic Blood Pressure and pulse wave velocity will be measured before dosing. Cardiovascular markers will be checked throughout the study. Patients will be monitored monthly after starting study treatment. Total treatment period: 4 months.
  Interventions: Drug: Paricalcitol; Drug: Ergocalciferol

INTERVENTIONS:
Drug: Paricalcitol — 1. Patients will receive 1mcg once daily orally if iPTH is less than 500pg/ml;
  2. Patients will receive 2mcg once daily orally if iPTH is more than 500pg/ml. Duration of administration will be 16 weeks.
Drug: Ergocalciferol — 1. If baseline 25 OHD level is less than 5ng/mml: ergocalciferol 50,000 units once a week orally for 12 weeks, then 50,000 units monthly for total duration of 16 weeks.
  2. If baseline 25 OHD is between 5 and 15mg/ml: Ergocalciferol 50,000 units once a week orally for 4 weeks, then 50,000 units once a month for total duration of 16 weeks.
  3. If baseline 25 OHD level is between 16 and 30ng/ml: Ergocalciferol 50,000 units orally once every 4 weeks for 16 weeks.

SUMMARY:
This is an open label, single center, randomized, active comparator controlled study, comparing the effects of vitamin D replacement using oral ergocalciferol versus paricalcitol on parathyroid hormone (PTH) levels in patients with stage 3 and 4 CKD and vitamin D deficiency or insufficiency. The purpose of this study is to determine which of these two approaches is more successful.

DETAILED DESCRIPTION:
This study will enroll chronic kidney disease patients, stage 3 and 4, who have low serum vitamin D levels as defined by K DOQI Guidelines. Patients will be randomized to receive oral daily ergocalciferol or paricalcitol. A total of 80 patients will be enrolled, 40 in the cholecalciferol group and 40 in the paricalcitol group. Outcomes will be assessed as proportion of patients achieving pre-defined changes from baseline and as absolute changes from baseline values. Baseline values will be determined from averaging two consecutive measurements of the variables of interest prior to randomization.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female chronic kidney disease patients at least 18 years of age.
2. Patients should be able and willing to provide written informed consent and HIPAA Authorization.
3. Chronic kidney disease stage 3 or 4.
4. Plasma intactPTH level above 75pg/ml.
5. Serum 25 OHD level below 30ng/ml.
6. Negative pregnancy test unless 2 years postmenopausal or with a documented tubal ligation or total hysterectomy.
7. Patients need to be off of any Vitamin analogues or preparations for 4 weeks prior to screening.

Exclusion Criteria:

1. Women who are breast feeding, pregnant, capable of becoming pregnant, and not participating in an acceptable form of birth control.
2. Patients currently participating in a clinical trial with another investigational drug or device or who have receive an investigational drug or device within 30 days of enrollment in this study.
3. Major surgery within one month prior to enrollment or planned surgery while patient is in study (other than dialysis vascular access surgery).
4. Patients who have had a malignancy unless they have received curative treatment and have been disease free for 2 years.
5. Patients with a medical status that the PI decides would preclude participation.
6. Patients on hemodialysis or peritoneal dialysis.
7. Patients with a functional renal transplant.
8. Patients with allergies to study drugs.
9. Patients with acute renal failure with the past 12 weeks.
10. Patients with clinically significant gastrointestinal or liver disease.
11. Patients with active granulomatous disease.
12. Patients with urine calcium:creatinine ratio of more than 0.2.
13. Patients who received vitamin D analogs, calcimimetics, or biphosphonates within 4 weeks before screening. Treatment with any one of these medicines during the study is not permitted.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2009-07; Primary Completion 2011-01 (Actual); Study Completion 2011-01 (Actual)

PRIMARY OUTCOMES:
To achieve 2 consecutive iPTH measurements with 30% or greater decrease from baseline | 2 years

SECONDARY OUTCOMES:
To achieve 25OHD level above 30 ng/ml and change cardiovascular markers | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Csaba P. Kovesdy, M.D., Principal Investigator — Salem VAMC
Locations (1):
- VA Medical Center, Salem, Virginia, United States